CLINICAL TRIAL: NCT00107315
Title: A Phase II Study of Capecitabine and Bevacizumab in Elderly Patients With Metastatic Colorectal Cancer
Brief Title: Bevacizumab and Capecitabine as First-Line Therapy in Treating Older Patients With Metastatic Colorectal Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Terminated due to low accrual
Sponsor: Roswell Park Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: I 22204; RPCI-I-22204; GENENTECH-RPCI-I-22204
Record Dates: First submitted 2005-04-05; First posted 2005-04-06 (Estimated); Results first posted 2014-07-04 (Estimated); Last update posted 2014-07-04 (Estimated); Status verified 2014-06

CONDITIONS: Colorectal Cancer
Keywords: recurrent colon cancer; stage IV colon cancer; recurrent rectal cancer; stage IV rectal cancer
MeSH Terms: conditions — Colorectal Neoplasms; Colonic Neoplasms; Rectal Neoplasms | interventions — Bevacizumab; Capecitabine

ARMS (1):
- Arm 1 (Experimental): Patients receive bevacizumab IV over 30-90 minutes on day 1 and oral capecitabine twice daily on days 1-7
  Interventions: Biological: bevacizumab; Drug: capecitabine

INTERVENTIONS:
Biological: bevacizumab
Drug: capecitabine

SUMMARY:
RATIONALE: Monoclonal antibodies, such as bevacizumab, can block tumor growth in different ways. Some block the ability of tumor cells to grow and spread. Others find tumor cells and help kill them or carry tumor-killing substances to them. Bevacizumab may also stop the growth of colorectal cancer by blocking blood flow to the tumor. Drugs used in chemotherapy, such as capecitabine, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving bevacizumab together with capecitabine may kill more tumor cells.

PURPOSE: This phase II trial is studying how well giving bevacizumab together with capecitabine works as first-line therapy in treating older patients with metastatic colorectal cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the time to disease progression in older patients with metastatic colorectal cancer treated with bevacizumab and capecitabine as first-line therapy.

Secondary

* Determine the response rate in patients treated with this regimen.
* Determine the median survival of patients treated with this regimen.
* Determine the toxic effects of this regimen in these patients.

OUTLINE: This is an open-label study.

Patients receive bevacizumab IV over 30-90 minutes on day 1 and oral capecitabine twice daily on days 1-7. Courses repeat every 14 days in the absence of disease progression or unacceptable toxicity.

PROJECTED ACCRUAL: A total of 40 patients will be accrued for this study within 13-16 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically* or cytologically* confirmed colorectal cancer

  * Site of primary tumor must have been confirmed by endoscopy, radiography, or surgery
  * Metastatic disease NOTE: *Patients with a history of surgically treated colorectal cancer who subsequently develop recurrent metastatic disease do not require histologic or cytologic confirmation of metastatic disease unless an interval of > 5 years has elapsed between initial primary surgery and the development of metastases
* Measurable disease

  * At least 1 unidimensionally measurable lesion ≥ 20 mm by conventional techniques OR ≥ 10 mm by spiral CT scan
* No known curative therapy exists
* No history or evidence of CNS disease by physical exam (e.g., primary brain tumor or brain or CNS metastases)

PATIENT CHARACTERISTICS:

Age

* 70 and over

Performance status

* ECOG 0-1

Life expectancy

* More than 3 months

Hematopoietic

* Absolute neutrophil count ≥ 1,500/mm^3
* Platelet count ≥ 100,000/mm^3
* Hemoglobin ≥ 9 g/dL
* No bleeding diathesis or coagulopathy

Hepatic

* Bilirubin normal
* AST and ALT ≤ 3 times upper limit of normal (ULN)
* INR < 1.5 (unless on therapeutic anticoagulants)
* No unstable or uncompensated hepatic disease

Renal

* Creatinine < 1.2 times ULN OR
* Creatinine clearance > 60 mL/min
* No unstable or uncompensated renal disease

Cardiovascular

* No history of stroke
* No uncontrolled hypertension (i.e., blood pressure > 150/100 mm Hg on medication)
* No myocardial infarction within the past year
* No New York Heart Association class II-IV congestive heart failure
* No unstable angina
* No serious cardiac dysrhythmia requiring medication
* No other clinically significant cardiovascular disease
* No other unstable or uncompensated cardiac disease

Pulmonary

* No unstable or uncompensated respiratory disease

Other

* Fertile patients must use effective contraception
* Able to receive oral medication
* No known hypersensitivity to fluorouracil or capecitabine
* No known dihydropyrimidine dehydrogenase deficiency
* No seizures not controlled by standard medical therapy
* No serious nonhealing wound, ulcer, or bone fracture
* No other malignancy within the past 5 years except completely excised nonmelanoma skin cancer (with no evidence of recurrent disease) or carcinoma in situ of the cervix
* No other severe or uncontrolled systemic disease

PRIOR CONCURRENT THERAPY:

Biologic therapy

* No prior bevacizumab

Chemotherapy

* Prior adjuvant fluorouracil and leucovorin calcium allowed provided the last treatment was administered > 6 months before the development of metastatic disease
* No prior chemotherapy for metastatic colon cancer
* No prior irinotecan or oxaliplatin

Endocrine therapy

* Not specified

Radiotherapy

* Not specified

Surgery

* See Disease Characteristics
* More than 28 days since prior and no concurrent major surgery
* More than 28 days since prior open biopsy
* More than 7 days since prior fine needle aspiration or core biopsy

Other

* More than 4 weeks since prior and no concurrent participation in another experimental drug study
* More than 30 days since prior non-approved or investigational drugs

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 16 (Actual)
Dates: Start 2004-07; Primary Completion 2008-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marwan Fakih, MD, Principal Investigator — Roswell Park Cancer Institute
Locations (1):
- Roswell Park Cancer Institute, Buffalo, New York, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Combination of Capecitabine and Bevacizumab: Patients received 1500 mg/m2/dose of capecitabine twice daily×7 days and bevacizumab at 5 mg/kg on day 1, in 2 week-cycles.
Period: Overall Study
Arm/Group | Combination of Capecitabine and Bevacizumab
Started | 16
Completed | 1
Not Completed | 15
Not completed — Disease Progression | 9
Not completed — Adverse Event | 4
Not completed — Withdrawal by Subject | 2

BASELINE CHARACTERISTICS:
Population: All treated and eligible patients
Arm/Group | Combination of Capecitabine and Bevacizumab
Number analyzed (Participants) | 16
Age, Continuous [Mean (Standard Deviation); unit: years] | 78 (4.9)
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 0
  >=65 years | 16
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 5

OUTCOME MEASURES:

1. Primary Outcome: Time to Progression
Time Frame: 1 year
Population: Due to the study's early termination and inadequate number of patients, no patients were analyzed.
Arm/Group | Combination of Capecitabine and Bevacizumab
Number analyzed (Participants) | 0

2. Secondary Outcome: Response Rate
Description: Overall Response (OR) = CR + PR.
Time Frame: 1 year
Population: Due to the study's early termination and inadequate number of patients, no patients were analyzed.
Arm/Group | Combination of Capecitabine and Bevacizumab
Number analyzed (Participants) | 0

3. Secondary Outcome: Median Survival
Time Frame: 1 year
Population: Due to the study's early termination and inadequate number of patients, no patients were analyzed.
Arm/Group | Combination of Capecitabine and Bevacizumab
Number analyzed (Participants) | 0

4. Secondary Outcome: Toxicity
Description: Number of participants with an adverse event.
  Please refer to the adverse event reporting for more detail.
Time Frame: 1 year
Population: Due to the study's early termination and inadequate number of patients, no patients were analyzed.
Arm/Group | Combination of Capecitabine and Bevacizumab
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | Combination of Capecitabine and Bevacizumab
Serious Adverse Events (participants affected / at risk) | 11/16
Other Adverse Events (participants affected / at risk) | 16/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Combination of Capecitabine and Bevacizumab (N=16)
Atrial thrombosis (Cardiac disorders) | 1 (2)
Diarrhoea (Gastrointestinal disorders) | 1 (2)
Enteritis (Gastrointestinal disorders) | 1 (1)
Intestinal ischaemia (Gastrointestinal disorders) | 1 (2)
Large intestine perforation (Gastrointestinal disorders) | 1 (2)
Nausea (Gastrointestinal disorders) | 1 (2)
Proctalgia (Gastrointestinal disorders) | 1 (2)
Vomiting (Gastrointestinal disorders) | 1 (2)
Pain (General disorders) | 1 (2)
Syncope (Nervous system disorders) | 1 (2)
Transient ischaemic attack (Nervous system disorders) | 2 (4)
Haematuria (Renal and urinary disorders) | 1 (2)
Pelvic pain (Reproductive system and breast disorders) | 1 (2)
Arterial thrombosis (Vascular disorders) | 1 (2)
Deep vein thrombosis (Vascular disorders) | 1 (2)
Venous thrombosis (Vascular disorders) | 1 (2)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Combination of Capecitabine and Bevacizumab (N=16)
Anaemia (Blood and lymphatic system disorders) | 4 (8)
Bradycardia (Cardiac disorders) | 1 (1)
Tinnitus (Ear and labyrinth disorders) | 1 (2)
Vertigo (Ear and labyrinth disorders) | 1 (2)
Dry eye (Eye disorders) | 1 (2)
Keratoconjunctivitis sicca (Eye disorders) | 1 (2)
Lacrimation increased (Eye disorders) | 1 (2)
Anal discomfort (Gastrointestinal disorders) | 1 (2)
Ascites (Gastrointestinal disorders) | 1 (2)
Diarrhoea (Gastrointestinal disorders) | 4 (17)
Dry mouth (Gastrointestinal disorders) | 1 (4)
Flatulence (Gastrointestinal disorders) | 1 (8)
Nausea (Gastrointestinal disorders) | 2 (3)
Stomatitis (Gastrointestinal disorders) | 3 (8)
Toothache (Gastrointestinal disorders) | 1 (2)
Vomiting (Gastrointestinal disorders) | 2 (4)
Chest pain (General disorders) | 1 (2)
Fatigue (General disorders) | 4 (9)
Injection site reaction (General disorders) | 2 (4)
Mucosal inflammation (General disorders) | 1 (1)
Oedema (General disorders) | 1 (6)
Oedema peripheral (General disorders) | 1 (2)
Pyrexia (General disorders) | 1 (2)
Hypersensitivity (Immune system disorders) | 1 (2)
Cystitis (Infections and infestations) | 1 (2)
Enteritis infectious (Infections and infestations) | 1 (2)
Nail infection (Infections and infestations) | 2 (4)
Nasopharyngitis (Infections and infestations) | 1 (2)
Pneumonia (Infections and infestations) | 1 (2)
Rhinitis (Infections and infestations) | 1 (4)
Sinusitis (Infections and infestations) | 1 (2)
Subcutaneous abscess (Infections and infestations) | 1 (2)
Upper respiratory tract infection (Infections and infestations) | 1 (2)
Urinary tract infection (Infections and infestations) | 2 (6)
Rib fracture (Injury, poisoning and procedural complications) | 1 (2)
Tooth injury (Injury, poisoning and procedural complications) | 1 (2)
Wound (Injury, poisoning and procedural complications) | 1 (2)
Alanine aminotransferase increased (Investigations) | 1 (4)
Aspartate aminotransferase increased (Investigations) | 1 (4)
Blood alkaline phosphatase increased (Investigations) | 1 (2)
Blood creatinine (Investigations) | 1 (2)
Haemoglobin (Investigations) | 1 (4)
Haemoglobin decreased (Investigations) | 1 (2)
Protein total increased (Investigations) | 1 (2)
Protein urine (Investigations) | 1 (2)
Weight increased (Investigations) | 1 (2)
Anorexia (Metabolism and nutrition disorders) | 2 (5)
Dehydration (Metabolism and nutrition disorders) | 2 (3)
Hyperglycaemia (Metabolism and nutrition disorders) | 8 (35)
Hyperkalaemia (Metabolism and nutrition disorders) | 2 (4)
Hypernatraemia (Metabolism and nutrition disorders) | 1 (2)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 3 (6)
Hypocalcaemia (Metabolism and nutrition disorders) | 2 (4)
Hypoglycaemia (Metabolism and nutrition disorders) | 2 (3)
Hypokalaemia (Metabolism and nutrition disorders) | 2 (3)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (4)
Convulsion (Nervous system disorders) | 1 (2)
Coordination abnormal (Nervous system disorders) | 2 (4)
Dizziness (Nervous system disorders) | 2 (4)
Dysgeusia (Nervous system disorders) | 1 (4)
Paraesthesia (Nervous system disorders) | 1 (4)
Depression (Psychiatric disorders) | 1 (2)
Cystitis-like symptom (Renal and urinary disorders) | 1 (2)
Dysuria (Renal and urinary disorders) | 1 (2)
Leukocyturia (Renal and urinary disorders) | 1 (2)
Stress urinary incontinence (Renal and urinary disorders) | 1 (2)
Urinary incontinence (Renal and urinary disorders) | 1 (2)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (4)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (8)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (2)
Blood blister (Skin and subcutaneous tissue disorders) | 1 (2)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (2)
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 14 (50)
Rash (Skin and subcutaneous tissue disorders) | 2 (4)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 1 (2)
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 (2)
Hypertension (Vascular disorders) | 4 (10)

LIMITATIONS AND CAVEATS:
Due to the study's early termination, as a result of low accrual, target accrual was not reached and no statistical inference of the primary and secondary aims were carried forth.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes